CLINICAL TRIAL: NCT01288924
Title: Can Preemptive Analgesia With Parecoxib Reduce Post-operative Ipsilateral Shoulder Pain? A Double-blinded, Randomized, Placebo-controlled Trial.
Brief Title: Can Parecoxib Reduce Post-operative Ipsilateral Shoulder Pain?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Tanyong Pipanmekaporn, Department of Anesthesiology,Faculty of Medicine, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: COM-10-11-19A-12; research ID 79 (Other: Ethic committee, Faculty of Medicine, Chiang Mai University)
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Shoulder Pain; Post-operative Pain
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative | interventions — parecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parecoxib (Active Comparator): Parecoxib 2 ml intravenous
  Interventions: Drug: Parecoxib
- Control (Placebo Comparator): 0.9% sodium chloride 2 ml intravenous
  Interventions: Other: Control

INTERVENTIONS:
Drug: Parecoxib — Parecoxib 40 mg intravenous before surgery and every 12 hours for two days.
  Other Names: Dynastat
  Arms: Parecoxib
Other: Control — NSS 2 ml intravenous before surgery and every 12 hours for two days.
  Arms: Control

SUMMARY:
The purpose of this study is to compare the efficacy of parecoxib with placebo on the incidence and severity of postthoracotomy shoulder pain, the amount of analgesic requirement for relieving severity of postthoracotomy shoulder pain and adverse events associated with treatment.

DETAILED DESCRIPTION:
The incidence of Post-operative Ipsilateral Shoulder Pain (PISP) varies from 21-97% after thoracic surgery, despite receiving effective thoracic epidural analgesia. This pain has been described as constant, aching in quality, unrelated to position change or respiration. Possible causes of shoulder pain includes injury of the phrenic nerve, the lateral decubitus position, transection of major bronchus or preexisting arthritis condition. The possibilities of prevention and management of PISP are taken into consideration. Thoracic epidural block will be performed in all patients before general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical status I-III
* Undergoing pulmonary resection by open thoracotomy

Exclusion Criteria:

* Unable to understand numeric rating scale despite preoperative coaching
* Preexisting shoulder pain at the same operative side
* Having contraindication for thoracic epidural analgesia
* History of previous myocardial ischemia or cerebrovascular accident
* Allergic to NSAIDS, sulfonamides or parecoxib
* Hepatic or renal impairment
* History of current gastrointestinal symptoms
* Fluid retention or congestive heart failure
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-02; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) of shoulder pain and incisional pain at rest and movement | at 2 ,6 ,12 ,24 ,48,72 and 96 hours after the operation

SECONDARY OUTCOMES:
compare an amount of morphine consumption | at 2,6 ,12,24,48,72 and 96 hours after the operation
adverse effect related to parecoxib | during 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tanyong Pipanmekaporn, MD, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Chiang Mai University , Chiang Mai, Thailand,50200
Locations (2):
- Thailand (2):
  - Department of Anesthesiology, Faculty of Medicine, Chiang Mai University, Maung, Chiang Mai
  - Department of Anesthesiology, Faculty of Medicine, Maung, Chiang Mai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bamgbade OA, Dorje P, Adhikary GS. The dual etiology of ipsilateral shoulder pain after thoracic surgery. J Clin Anesth. 2007 Jun;19(4):296-8. doi: 10.1016/j.jclinane.2006.09.010. PMID 17572327
- [Background] MacDougall P. Postthoracotomy shoulder pain: diagnosis and management. Curr Opin Anaesthesiol. 2008 Feb;21(1):12-5. doi: 10.1097/ACO.0b013e3282f2bb67. PMID 18195603